CLINICAL TRIAL: NCT00000914
Title: A Randomized Study of the Virologic Efficacy of Different Antiretroviral (AR) Treatment Strategies in HIV-Infected Individuals With Detectable Plasma HIV RNA Measurements After at Least 16 Weeks on Their Initial Protease Inhibitor-Containing AR Regimens
Brief Title: A Study of the Effectiveness of Different Anti-HIV Treatments in HIV-Positive Individuals Who Have Been on a Protease Inhibitor-Containing Drug Regimen for at Least 16 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CPCRA 057; 11610 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; Saquinavir; Reverse Transcriptase Inhibitors; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Nelfinavir; efavirenz

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Efavirenz

SUMMARY:
The purpose of this study is to compare different treatments for HIV infection to see which works best to lower HIV levels and to raise the number of CD4 cells (cells of the immune system that fight infection), in HIV-positive individuals who have been on a protease inhibitor-containing drug regimen for at least 16 weeks.

Researchers have found that combination anti-HIV therapy (multiple drugs given together) can help prevent AIDS-related illnesses and help people with AIDS live longer. In this study, the anti-HIV drug efavirenz (EFV) will be tested with 1 or 2 other protease inhibitors (PIs) to see which combination works best to treat HIV infection. EFV has been shown to limit the amount of HIV virus produced by infected cells.

DETAILED DESCRIPTION:
Current recommendations for the initial treatment of HIV infection have centered on the reduction of plasma HIV levels. It has been shown that a combination of 2 nucleoside reverse transcriptase inhibitors (NRTIs) and a PI is the most effective barriers to disease progression. This study attempts to demonstrate these data.

Two options are available for patients whose initial PI-containing regimen has failed to suppress viral replication.

Option 1 consists of immediate versus deferred use of a nonnucleoside reverse transcriptase inhibitor (NNRTI). Patients who choose Option 1 are randomized to 1 of 2 groups:

1. Ritonavir (RTV) plus soft gelatin capsule saquinavir (SQV-SGC) plus efavirenz (EFV).
2. RTV plus SQV-SGC.

Option 2 consists of treatment with a single PI versus double PI. Patients who choose Option 2 are randomized to 1 of 2 groups:

1. Nelfinavir (NFV) plus EFV.
2. RTV plus SQV-SGC plus EFV.

Patients failing NFV in Option 2 are randomized to one of two groups:

1. Indinavir (IDV) plus EFV.
2. RTV plus SQV-SGC plus EFV. Patients remain on study treatment regimens for 8 weeks. Follow-up visits, including history and physical evaluations, take place at specified intervals during the next 12 months.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have an HIV RNA count of at least 400 copies/ml.
* Are at least 13 years old (need consent if under 18).
* Have been on antiretroviral treatment (including at least 2 NRTIs) for at least 16 weeks prior to study entry.
* Agree to practice abstinence or to use effective methods of birth control, including a barrier method, during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Are pregnant or breast-feeding.
* Have active opportunistic (HIV-associated) infections.
* Have taken nelfinavir (NFV) for more than 2 weeks after failing indinavir/ritonavir (IDV/RTV) treatment or have taken IDV/RTV for more than 2 weeks after failing NFV treatment.
* Have used any protease inhibitor other than NFV or IDV/RTV for more than 2 weeks.
* Have used any non-nucleoside reverse transcriptase inhibitor (NNRTI) for more than 1 week.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay R. Kostman, Study Chair; Lawrence R. Crane, Study Chair
Locations (15):
- United States (15):
  - Community Consortium / UCSF, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Washington Reg AIDS Prog / Dept of Infect Dis, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ - WSU/DMC / Univ Hlth Ctr, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Harlem AIDS Treatment Grp / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium / Div of Infect Diseases, Richmond, Virginia

REFERENCES:
- [Background] Mannheimer S, Friedland G, Matts J, Child C, Chesney M. Antiretroviral adherence correlates with quality of life. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 485)